CLINICAL TRIAL: NCT03302130
Title: The Effects of Mood on Cerebral Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC/2015/0528
Record Dates: First submitted 2016-10-06; First posted 2017-10-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Perfusion
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging healthy volunteers (Experimental): Mood induction: positive, negative, neutral mood (using subjects own memories) Arterial spin labeling MRI Physiological monitoring
  Interventions: Behavioral: Mood induction (using own memories); Device: Arterial spin labeling MRI; Device: Physiological monitoring

INTERVENTIONS:
Behavioral: Mood induction (using own memories) — Subjects deliver three positive, three negative and three neutral memories 30 seconds reliving a memory - answering questions about the memory - reliving memory for 2 minutes during ASL-MRI
Device: Arterial spin labeling MRI — Single PLD PCASL
Device: Physiological monitoring — During MRI: heart rate, end-tidal CO2, respiratory rate and skin conductance

SUMMARY:
Measuring brain perfusion is biased by a inter- and intrasubject variability, caused by physiological and lifestyle factors. In this study, the investigators want to investigate the effects of a different mood state (neutral, positive and negative mood), induced using subjects own memories, on both global and regional cerebral perfusion, measured with arterial spin labeling.

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students
* between 18 and 30 years old

Exclusion Criteria:

* No informed consent
* Not using hormonal contraception
* MRI-contraindications
* Claustrophobia
* Pregnancy
* Chronic diseases and chronic medication use

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Regional Cerebral perfusion (ml/100g/min) during positive mood induction | 2 minutes (ASL scan during mood state induction)
  Effect of positive mood induction (using volunteer's own memories) on cerebral perfusion using arterial spin labeling MRI.
Regional Cerebral perfusion (ml/100g/min) during negative mood induction | 2 minutes (ASL scan during mood state induction)
  Effect of negative mood induction (using volunteer's own memories) on cerebral perfusion using arterial spin labeling MRI.
Regional Cerebral perfusion (ml/100g/min) during neutral mood induction | 2 minutes (ASL scan during mood state induction)
  Effect of neutral mood induction (using volunteer's own memories) on cerebral perfusion using arterial spin labeling MRI.
Regional Cerebral perfusion (ml/100g/min) after positive mood induction | 2 minutes (ASL scan after mood state induction)
  Effect of positive mood (using volunteer's own memories) on cerebral perfusion using arterial spin labeling MRI.
Regional Cerebral perfusion (ml/100g/min) after negative mood induction | 2 minutes (ASL scan after mood state induction)
  Effect of negative mood (using volunteer's own memories) on cerebral perfusion using arterial spin labeling MRI.
Regional Cerebral perfusion (ml/100g/min) after neutral mood induction | 2 minutes (ASL scan after mood state induction)
  Effect of neutral mood (using volunteer's own memories) on cerebral perfusion using arterial spin labeling MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Achten, MD, PhD, Principal Investigator — University Hospital, Ghent